CLINICAL TRIAL: NCT00026559
Title: Effects of Arousal and Stress on Classical Conditioning
Brief Title: Effects of Arousal and Stress in Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 010185; 01-M-0185
Record Dates: First submitted 2001-11-10; First posted 2001-11-12 (Estimated); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2022-07-28

CONDITIONS: Healthy Volunteers
Keywords: Classical Conditioning; Fear Conditioning; Stress; Learning; Normal Volunteers; Healthy Volunteer; Normal Control

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Healthy volunteers (Experimental): Sub-study A: Working memory task / Participant performed a working memory task in two conditions, under threat of shock and in safety and asked to remember verbal and nonverbal stimuli from the current stimulus on the screen (N-back task) Sub-study C: Sustained attention to response task (SART) / participant was presented with stimuli and either initiated a response (i.e. "go") or inhibited their response (i.e. "stop") based on what stimuli were presented Sub-study D: Stroop task/ In the classic Stroop test, the name of a color is printed in a color that conflicts or does not conflict with the word. In the emotional Stroop, the words emotional words. The participant's task was to name the color of the word Pilot studies / (1) Shocks were delivered via electrodes located on the forearm or fingers while participant performed a working memory or vigilance task or (2) Subject performed cognitive tasks during alternating safe and threat periods
  Interventions: Device: Shock Device; Device: Auditory Startle Device

INTERVENTIONS:
Device: Shock Device — Shock Device
Device: Auditory Startle Device — Auditory Startle Device

SUMMARY:
This study has several parts. One part will examine the influence of factors such as personality and past experience on reactions to unpleasant stimuli. Others will examine the effect of personality and emotional and attentional states on learning and memory.

When confronted with fearful or unpleasant events, people can develop fear of specific cues that were associated with these events as well as to the environmental context in which the events occurred via a process called classical conditioning. Classical conditioning has been used to model anxiety disorders, but the relationship between stress and anxiety and conditioned responses remains unclear. This study will examine the relationship between cued conditioning and context conditioning . This study will also explore the acquisition and retention of different types of motor, emotional, and cognitive associative processes during various tasks that range from mildly arousing to stressful.

DETAILED DESCRIPTION:
Objective: Fear and anxiety are adaptive responses to different types of threats. Fear is a short-duration response evoked by explicit threat cues and anxiety a more sustained state of apprehension evoked by unpredictable threat. This protocol studied fear using Pavlovian fear conditioning in two studies. Studies 1 and 3. Study 2 focused on anxiety. Studies 1 and 3 will be discontinued to focus uniquely on the study of anxiety. Specifically, we will examine the interactions between anxiety induced experimentally using verbal threat and cognitive processes. We will seek to 1) characterize the effect of anxiety on key cognitive processes including working memory and attention control and 2) examine the extent to which performance of cognitive tasks distract from anxiety.

Study population: This more-than-minimal-risk protocol will test medically and psychiatrically healthy volunteers aged 18-50. Pregnant or nursing women will be excluded.

Method: Fear and anxiety will be measured using the startle reflex to brief and loud sounds. Fear conditioning will be assessed using shock as unconditioned stimulus. Cognitive performance will be examined during periods of unpredictable shock anticipation.

Outcome measures: The study will include cognitive performance and measure of aversive states, primarily the startle reflex.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Males and females
* Age 18-50

EXCLUSION CRITERIA:

* Pregnancy
* Any current ongoing medical illness
* Current Axis I disorders
* Past significant psychiatric disorders (e.g., psychotic disorders) according to Diagnostic and Statistical Manual (DSM)-IV
* Current alcohol or substance abuse according to DSM-IV criteria
* History of alcohol or substance dependence based on DSM-IV criteria within 6 months prior to screening
* Current psychotropic medication use
* Current or past organic central nervous system disorders, including but not limited to seizure disorder or neurological symptoms of the wrist and arms (e.g., carpal tunnel syndrome). The latter exclusion is for shock studies only.
* Positive urine toxicology screen
* Employees of National Institute of Mental Health (NIMH) or an immediate family member of a NIMH employee.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1418 (Actual)
Dates: Start 2001-01-10 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryland Pao, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We will provide de-identified data to repositories but no identifiable data.

REFERENCES:
- [Background] Grillon C, Morgan CA 3rd. Fear-potentiated startle conditioning to explicit and contextual cues in Gulf War veterans with posttraumatic stress disorder. J Abnorm Psychol. 1999 Feb;108(1):134-42. doi: 10.1037//0021-843x.108.1.134. PMID 10066999
- [Background] Grillon C, Ameli R, Goddard A, Woods SW, Davis M. Baseline and fear-potentiated startle in panic disorder patients. Biol Psychiatry. 1994 Apr 1;35(7):431-9. doi: 10.1016/0006-3223(94)90040-x. PMID 8018793
- [Background] Phillips RG, LeDoux JE. Differential contribution of amygdala and hippocampus to cued and contextual fear conditioning. Behav Neurosci. 1992 Apr;106(2):274-85. doi: 10.1037//0735-7044.106.2.274. PMID 1590953
- [Result] Balderston NL, Liu J, Roberson-Nay R, Ernst M, Grillon C. The relationship between dlPFC activity during unpredictable threat and CO2-induced panic symptoms. Transl Psychiatry. 2017 Nov 30;7(12):1266. doi: 10.1038/s41398-017-0006-5. PMID 29213110
- [Result] Grillon C, Robinson OJ, Krimsky M, O'Connell K, Alvarez G, Ernst M. Anxiety-mediated facilitation of behavioral inhibition: Threat processing and defensive reactivity during a go/no-go task. Emotion. 2017 Mar;17(2):259-266. doi: 10.1037/emo0000214. Epub 2016 Sep 19. PMID 27642657
- [Result] Grillon C, Robinson OJ, Mathur A, Ernst M. Effect of attention control on sustained attention during induced anxiety. Cogn Emot. 2016;30(4):700-12. doi: 10.1080/02699931.2015.1024614. Epub 2015 Apr 22. PMID 25899613
- [Result] Lago TR, Hsiung A, Leitner BP, Duckworth CJ, Balderston NL, Chen KY, Grillon C, Ernst M. Exercise modulates the interaction between cognition and anxiety in humans. Cogn Emot. 2019 Jun;33(4):863-870. doi: 10.1080/02699931.2018.1500445. Epub 2018 Jul 23. PMID 30032703
- [Derived] Roxburgh AD, White DJ, Grillon C, Cornwell BR. A neural oscillatory signature of sustained anxiety. Cogn Affect Behav Neurosci. 2023 Dec;23(6):1534-1544. doi: 10.3758/s13415-023-01132-1. Epub 2023 Oct 25. PMID 37880568
- [Derived] Grillon C, Ernst M. A way forward for anxiolytic drug development: Testing candidate anxiolytics with anxiety-potentiated startle in healthy humans. Neurosci Biobehav Rev. 2020 Dec;119:348-354. doi: 10.1016/j.neubiorev.2020.09.024. Epub 2020 Oct 7. PMID 33038346
- [Derived] Grillon C, Lago T, Stahl S, Beale A, Balderston N, Ernst M. Better cognitive efficiency is associated with increased experimental anxiety. Psychophysiology. 2020 Aug;57(8):e13559. doi: 10.1111/psyp.13559. Epub 2020 Mar 17. PMID 32180239
- [Derived] Sarigiannidis I, Grillon C, Ernst M, Roiser JP, Robinson OJ. Anxiety makes time pass quicker while fear has no effect. Cognition. 2020 Apr;197:104116. doi: 10.1016/j.cognition.2019.104116. Epub 2019 Dec 26. PMID 31883966
- [Derived] Robinson OJ, Pike AC, Cornwell B, Grillon C. The translational neural circuitry of anxiety. J Neurol Neurosurg Psychiatry. 2019 Dec;90(12):1353-1360. doi: 10.1136/jnnp-2019-321400. Epub 2019 Jun 29. PMID 31256001
- [Derived] Balderston NL, Hsiung A, Liu J, Ernst M, Grillon C. Reducing State Anxiety Using Working Memory Maintenance. J Vis Exp. 2017 Jul 19;(125):55727. doi: 10.3791/55727. PMID 28745646
- [Derived] Lago T, Davis A, Grillon C, Ernst M. Striatum on the anxiety map: Small detours into adolescence. Brain Res. 2017 Jan 1;1654(Pt B):177-184. doi: 10.1016/j.brainres.2016.06.006. Epub 2016 Jun 6. PMID 27276526
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-M-0185.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All sub-studies were conducted at different time points so subjects had the option to participate in multiple sub-studies
Groups:
- Healthy Volunteers: Healthy volunteers participated in one or more sub-studies:
  Sub-study A: Working memory and anxiety / Participant performed a working memory task in two conditions, under threat of shock and in safety and asked to remember verbal and nonverbal stimuli from the current stimulus on the screen (N-back task).
  Sub-study C: Effect of anxiety on sustained attention to response task (SART) / participant was presented with stimuli and either initiated a response (i.e. "go") or inhibited their response (i.e. "stop") based on what stimuli were presented.
  Sub-study D: Effect of anxiety on Stroop task/ In the classic Stroop test, the name of a color is printed in a color that conflicts or does not conflict with the word. In the emotional Stroop, the words emotional words. The participant's task was to name the color of the word.
  Pilot studies / (1) Shocks were delivered via electrodes located on the forearm or fingers while participant performed a working memory or vigilance task or (2) Subject performed cognitive tasks during alternating safe and threat periods
Period: Healthy Volunteers
Arm/Group | Healthy Volunteers
Started | 1418
Completed | 1418
Not Completed | 0
Period: Working Memory Task
Arm/Group | Healthy Volunteers
Started | 115
Completed | 115
Not Completed | 0
Period: Sustained Attention to Response Task
Arm/Group | Healthy Volunteers
Started | 61 (Include seven subjects who also participated in the working memory task sub-study)
Completed | 61
Not Completed | 0
Period: Stroop Task
Arm/Group | Healthy Volunteers
Started | 69 (Include 28 subjects who also participated in the working memory task and two subjects who participated in the Sustained attention to response task sub-studies)
Completed | 69
Not Completed | 0
Period: Pilot Studies
Arm/Group | Healthy Volunteers
Started | 1210
Completed | 1210
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sub-study A: Working Memory Task: Participant performed a working memory task in two conditions, under threat of shock and in safety and asked to remember verbal and nonverbal stimuli from the current stimulus on the screen (N-back task)
- Sub-study C: Sustained Attention to Response Task (SART): Participant was presented with stimuli and either initiated a response (i.e. "go") or inhibited their response (i.e. "stop") based on what stimuli were presented
- Sub-study D: Stroop Task: In the classic Stroop test, the name of a color is printed in a color that conflicts or does not conflict with the word. In the emotional Stroop, the words emotional words. The participant's task was to name the color of the word
- Pilot Studies: (1) Shocks were delivered via electrodes located on the forearm or fingers while participant performed a working memory or vigilance task or (2) Subject performed cognitive tasks during alternating safe and threat periods
- Total: Total of all reporting groups
Arm/Group | Sub-study A: Working Memory Task | Sub-study C: Sustained Attention to Response Task (SART) | Sub-study D: Stroop Task | Pilot Studies | Total
Number analyzed (Participants) | 115 | 54 | 39 | 1210 | 1418
Age, Categorical [Count of Participants; unit: Participants]
  Healthy volunteers: <=18 years | 0 | 0 | 0 | 0 | 0
  Healthy volunteers: Between 18 and 65 years | 115 | 54 | 39 | 1210 | 1418
  Healthy volunteers: >=65 years | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Healthy volunteers: Female | 68 | 38 | 26 | 655 | 787
  Healthy volunteers: Male | 47 | 16 | 13 | 554 | 630
  Healthy volunteers: Unknown | 0 | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Healthy volunteers: Hispanic or Latino | 12 | 4 | 1 | 89 | 106
  Healthy volunteers: Not Hispanic or Latino | 101 | 48 | 38 | 1103 | 1290
  Healthy volunteers: Unknown or Not Reported | 2 | 2 | 0 | 18 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Healthy volunteers: American Indian or Alaska Native | 0 | 0 | 0 | 7 | 7
  Healthy volunteers: Asian | 22 | 7 | 3 | 169 | 201
  Healthy volunteers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 3 | 3
  Healthy volunteers: Black or African American | 26 | 20 | 13 | 280 | 339
  Healthy volunteers: White | 58 | 23 | 21 | 662 | 764
  Healthy volunteers: More than one race | 6 | 1 | 1 | 26 | 34
  Healthy volunteers: Unknown or Not Reported | 3 | 3 | 1 | 63 | 70

OUTCOME MEASURES:

1. Primary Outcome: Go Correct Hits Followed by Button Press
Description: Subjects participated in go/no go (GNG) task condition during periods of threat of shocks and periods of safety when no shock could be administered. During the GNG stimuli were presented on a monitor. In the GNG task, participants were asked to respond to frequent 'go' stimuli ('=') by pressing the '2' on the keypad of a computer keyboard and to withhold their response to infrequent 'nogo' stimuli ('O'). Stimuli were randomly distributed. A correct go hit was a response recorded during these 2000 millisecond (ms) to a go trial. Similarly, a correct nogo omission was a no response during the same period to a nogo trial. Performance was determined for each condition (threat, safe) and trial type (go, nogo) by dividing the number of correct response by the total number of each trial type.
Time Frame: 250 ms at a rate of one every 2000 ms
Population: Analysis included a subset of 40 health volunteers who participated in a study to examine the effect of anxiety induced by the threat of shock on Go/NoGo performance. Four subjects were excluded in the final analysis.
Measure: Mean (95% Confidence Interval); unit: Percentage of correct responses
Groups:
- Healthy Volunteers: Healthy subjects will perform a variety of cognitive tasks during alternating safe and threat periods. Occasional startle stimuli will be delivered to assess anxiety.
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
Percentage of correct responses
  Safe Condition | 90.9 [88.6 to 93.1]
  Threat Condition | 91.6 [89.2 to 94]

2. Primary Outcome: Nogo Trials Followed by no Button Press
Description: as for outcome 1
Time Frame: 250 ms at a rate of one every 2000 ms
Population: Analysis included a subset of 40 health volunteers who participated in a study to examine the effect of anxiety induced by the threat of shock on Go-NoGo performance. Four subjects were excluded in the final analysis
Measure: Mean (95% Confidence Interval); unit: Percentage of correct responses
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
Percentage of correct responses
  Safe Condition | 74.4 [70.8 to 78.6]
  Threat Condition | 81.2 [76.7 to 85.7]

3. Primary Outcome: Correct-go Reaction Time (RT)
Description: Correct go responses were go trials followed by button press. Mean reaction time (RT) was calculated for correct-go to evaluate speed-accuracy trade-off.
Time Frame: 2000 ms during trial
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: millisecond
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
millisecond
  Safe Condition | 358.5 [339.1 to 377.9]
  Threat Condition | 349.3 [331 to 367.5]

4. Primary Outcome: Response to Startle Reflex
Description: The startle reflex was elicited with a 103-decibel (dB) white noise (40-ms duration) delivered via headphone. The eyeblink component of the startle reflex was recorded binaurally with two AgCl electrodes placed under the left eye. The peak startle/eyeblink reflex magnitude was determined in the 20-100 ms timeframe. The shock was administered either on the left wrist or on the left middle and ring fingers, depending on where the desired intensity was reached. Startle stimuli were delivered between two go trials and go trials that followed a startle stimulus were not included in the analysis. A shock was delivered in two of the four threat blocks in each sequence, just prior to the last go trial, which was not included in the analysis (for a total of 4 shocks). Shock could be administered only in the threat condition and never in the safe condition. The results were analyzed using a Condition (safe, threat) x Task (task, no task) repeated ANOVA.
Time Frame: 20-100 ms window following the onset of the startle stimulus
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
milliseconds
  No Task - Safe condition | 44.2 [41.9 to 46.4]
  No Task - Threat condition | 57.5 [55 to 59.5]
  Task - Safe condition | 42.4 [41 to 43.9]
  Task - Threat condition | 53 [50.4 to 55.5]

5. Primary Outcome: Subjective Measures of Level of Anxiety
Description: Subjects retrospectively rated their level of anxiety using a scale of 1-10 where 1 = "not at all anxious" and 10 = "extremely anxious" at the end of each block of a sequence for a total of eight blocks. A block was defined as a combination of a condition (safe or threat) and a task (task or no task). The results were analyzed using a Condition (safe, threat) x Task (task, no task) repeated ANOVA.
Time Frame: Every 100 sec repeated 8 times
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
Units on a scale
  No Task - Safe Condition | 1.6 [1.2 to 1.8]
  No Task - Threat Condition | 3.4 [2.7 to 4.2]
  Task - Safe Condition | 1.6 [1.4 to 1.9]
  Task - Threat Condition | 3.6 [2.9 to 4.3]

6. Secondary Outcome: Measure of Attention Control
Description: Subjects completed the Attention Control Scale (ACS) prior to start of the study. The ACS is a 20-item self-report scale that measures attentional focusing (9 items) and attentional shifting (11 items) rated on a four-point likert scale from "1 - almost never" to "4 - always" with total score range of 20 to 80. Higher score on ACS reflect better ability to direct and maintain attention.
Time Frame: 1-3 weeks before start of study
Population: Analysis included a subset of 60 health volunteers who participated in a study to examine the effect of anxiety induced by threat of shock on the Sustained Attention to Response Task (SART).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 60
Units on a scale | 59.9 (0.9)

7. Secondary Outcome: Measure of Level of Anxiety
Description: The level of anxiety was assessed using the Trait Anxiety Inventory questionnaire. The Trait Anxiety Scale (T-Anxiety) evaluates relatively stable aspects of "anxiety proneness", including general states of calmness, confidence, and security. The Trait Anxiety Scale has 20 items. All items are rated on a 4-point scale: 1 = almost never, 2 = sometimes, 3 = often, and 4 = almost always.. The scale has a minimum score of 20 and a maximum score of 80. Higher score indicates greater anxiety. Trait Anxiety score was measured prior to start of the study.
Time Frame: 1-3 weeks before start of study
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 60
Units on a scale | 28 (0.8)

ADVERSE EVENTS:
Time Frame: Up to four hours in a single day visit
Arm/Group | Sub-study A: Working Memory Task | Sub-study C: Sustained Attention to Response Task (SART) | Sub-study D: Stroop Task | Pilot Studies
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/61 | 0/69 | 0/1210
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/61 | 0/69 | 0/1210
Other Adverse Events (participants affected / at risk) | 0/115 | 0/61 | 0/69 | 0/1210

LIMITATIONS AND CAVEATS:
This protocol was a series of sub-studies using sample subjects which explains the low numbers of participants per study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT00026559/Prot_SAP_000.pdf